CLINICAL TRIAL: NCT04297072
Title: Adverse ReNal OuTcomEs in Patients With NoN-Valvular Atrial Fibrillation Treated With Rivaroxaban or Vitamin K Antagonists
Brief Title: Study to Gather Information on the Kidney Function of Patients With Non-valvular Atrial Fibrillation (Irregularly Heart Beats Which is Not Caused by a Heart Valve Problem) Treated With Rivaroxaban or Vitamin K Antagonists
Acronym: ANTENNA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 21347
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Non-Valvular Atrial Fibrillation
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rivaroxaban: Participants in this group administered oral anticoagulant Rivaroxaban
  Interventions: Drug: Rivaroxaban (Xarelto, BAY-597939)
- Vitamin-K antagonists (VKAs): Participants in this group administered oral anticoagulants VKAs
  Interventions: Drug: VKAs

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY-597939) — Non-vitamin K antagonist oral anticoagulants (NOACs). The prescription of drug is at the discretion of physician following the routine clinical practice.
  Groups: Rivaroxaban
Drug: VKAs — Oral anticoagulant. The prescription of drug is at the discretion of physician following the routine clinical practice.
  Groups: Vitamin-K antagonists (VKAs)

SUMMARY:
By evaluating routine clinical practice data from the UK primary care database, researchers in this study want to gather information on the kidney function of patients with non-valvular atrial fibrillation (NVAF, irregularly heart beats which is not caused by a heart valve problem) who are treated with Rivaroxaban (non-vitamin K antagonist, brand name Xarelto) or vitamin K antagonists (VKAs). The study planned to enroll about 25,000 male or female patients who were at least 18 years old and were new users of Rivaroxaban or VKAs between 01 January 2014 and 30 September 2019. Researchers are especially interested in whether patients experienced under treatment any worsening in kidney function, the onset of acute kidney diseases or injuries. In addition, risk of worsening in kidney function in patients with or without diabetes or heart failures are of interest to the researchers.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years in the IMRD-UK database
* a first prescription for either rivaroxaban or a VKA between 01 January 2014 and 31 March 2019. The date of the first rivaroxaban/VKA prescription will be set as the start date (start of follow-up for that patient). The follow-up will be extended until 30 September 2019 to ensure that each patient has at least 6 months of potential follow-up.
* a diagnosis of AF recorded any time before start date or within 2 weeks after start date.
* registered with their general practice at least 1 year before the start date and have a recorded prescription of any drug at least 1 year before the start date.
* registered with a general practice with data considered to be up-to-standard quality.

Exclusion Criteria:

* a prescription for any OAC before the start date - all first-time rivaroxaban/VKA users will therefore be OAC naïve
* a record of heart valve replacement or mitral stenosis any time before the start date or in the 2 weeks after the start date.
* a record of deep vein thrombosis, pulmonary embolism, or hip/knee surgery in the 3 months before the start date (because these are all alternative reasons for NOAC initiation).
* a record of ESRD (including renal transplant patients) on/before the start date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years with NVAF and no record of ESRD, with a first prescription for rivaroxaban or a VKA and no previous OAC use between 01 January 2014 and 30 September 2019
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
A 20%, 30%, 40%, or 50% increase in serum creatinine (SCr) at any point of time during follow-up (confirmed by a subsequent measurement) | Retrospectively analysis from 01 January 2014 to 30 September 2019
Doubling of SCr from initiation (start date) at any point of time during follow-up | Retrospectively analysis from 01 January 2014 to 30 September 2019
Rate of change in eGFR from initiation (start date) | Retrospectively analysis from 01 January 2014 to 30 September 2019
  To be included in the estimated glomerular filtration rates (eGFR) slope analyses at least two post-baseline assessments were required, where the first measurement was less than 120 days after index and the last was more than 180 days after the first post-baseline (reflecting sufficient time for a potential change to occur)
A 20%, 30%, 40%, or 50% decline of eGFR at any point of time during follow-up (confirmed by a subsequent measurement) | Retrospectively analysis from 01 January 2014 to 30 September 2019
Incidence of end-stage renal disease | Retrospectively analysis from 01 January 2014 to 30 September 2019
Incidence of acute kidney injury | Retrospectively analysis from 01 January 2014 to 30 September 2019

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.